CLINICAL TRIAL: NCT02231632
Title: Phase 2/3 Clinical Trial to Assess the Safety and Immunogenicity of Live Attenuated Poliomyelitis Vaccine (Human Diploid Cell)
Brief Title: The Immunogenicity and Safety of Live Attenuated Poliomyelitis Vaccine (Human Diploid Cell)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Yangjingsi2014
Record Dates: First submitted 2014-08-01; First posted 2014-09-04 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Poliomyelitis
Keywords: Poliomyelitis; Vaccine; Safety; efficacy
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Live attenuated Poliomyelitis vaccine (human diploid cell) (Experimental): 6.15 lgCCID50(containing typeⅠattenuated poliomyelitis not lower than 6.0 lgCCID50，typeⅡnot lower than 5.0 lgCCID50，type Ⅲ not lower than 5.5 lgCCID50).
  Interventions: Biological: Live attenuated Poliomyelitis vaccine (Human Diploid Cell)
- Poliomyelitis（Live）Vaccine(Monkey Kidney Cell),Oral (Experimental): 6.15 lgCCID50(containing typeⅠattenuated poliomyelitis not lower than 6.0 lgCCID50，typeⅡnot lower than 5.0 lgCCID50，type Ⅲ not lower than 5.5 lgCCID50).
  Interventions: Biological: Live attenuated Poliomyelitis vaccine (Monkey Kidney Cell)

INTERVENTIONS:
Biological: Live attenuated Poliomyelitis vaccine (Human Diploid Cell) — 6.15 lgCCID50 /Vial, 0.1ml/dose(10 dose /Vial) in babies aged 2-3 months, three dose(4 weeks'interval for each Intervention).
  Other Names: Poliomyelitis（Live）Vaccine(Human Diploid Cell),Oral
  Arms: Live attenuated Poliomyelitis vaccine (human diploid cell)
Biological: Live attenuated Poliomyelitis vaccine (Monkey Kidney Cell) — 6.15 lgCCID50 /Vial, 0.1ml/dose(10 dose /Vial) in babies aged 2-3 months, three dose(4 weeks'interval for each Intervention).
  Other Names: Poliomyelitis（Live）Vaccine(Monkey Kidney Cell),Oral
  Arms: Poliomyelitis（Live）Vaccine(Monkey Kidney Cell),Oral

SUMMARY:
The purpose of this Phase 2/3 trial is to assess the safety and immunogenicity of Live attenuated Poliomyelitis vaccine (human diploid cell)

DETAILED DESCRIPTION:
Live attenuated Poliomyelitis vaccine (human diploid cell) is used for poliovirus prevention in children above 2 years old , Which was developed by Institute of Medical Biology , Chinese Academy of Medical Sciences , based on the other two products : Poliomyelitis Vaccine in Dragee Candy (Monkey Kidney Cell), Live ; and Poliomyelitis（Live）Vaccine (Monkey Kidney Cell),Oral . After its safety been proved in phase 1 clinical trail evaluation , the phase 2/3 trail was started in Guangxi Province, China during 2011-2012. The purpose of this trial is to assess the safety and immunogenicity in healthy children of 2,3 and 4 months old .

ELIGIBILITY:
Inclusion Criteria:Only subjects fulfilling all of the following criteria will be eligible for the study:

* People aged from 2 months to 4 months old.
* The subjects or subjects' guardians are able to understand and sign the informed consent
* The subjects or subjects' guardians allow to comply with the requirements of the protocol
* Subjects with temperature <=37.0°C on axillary setting
* The subjects have signed informed consent already

Exclusion Criteria:The subjects have never been vaccinated with any Poliomyelitis Vaccine.

-

Ages: 2 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Comparison of virogene VP1 genovariation between vaccinal I-III Sabin strains and poliovirus separated from faeces of study objects after vaccinated | up to 90 days
  20 children aged 4 years old and 20 infants aged 2 months were vaccinated with 3 dose of Live attenuated Poliomyelitis vaccine (human diploid cell). Their faeces on day 0,7,30,60 and 90 were collected and incubated in L20B and RD cells for 2 generations, in order to separate and amplify poliovirus I-III Sabin strains in faeces of study objects . Extract total viral RNA from the culture supernatants and detect virogene VP1 through RT-PCR and sequencing ,in order to test the genovariation of vaccinal I-III Sabin strains in faeces after vaccinated .

SECONDARY OUTCOMES:
The frequency of all the adverse events in vaccine group and placebo group | up to 30 days
  compare frequency of all the solicited events, unsolicited adverse events and serious adverse events between vaccine groups.
Change of seroconversion from baseline to 3 months | up to 3 months
  Randomly chose 600 infants respectively from two study arms, get 2.5ml of the blood on the first day and 3 months during vaccination .Reciprocal antibody titers of at least 1:8, the lowest detectable titer, is considered to indicate seropositivity with regards to the presence of poliovirus neutralizing antibodies. Seroconversion is defined as either seronegative participants (<1:8 titers) who become seropositive (≥1:8) or participants who demonstrate a 4-fold change in titers between two specimens, e.g. a change from 1:8 to 1:32. Chi-square tests will be used to test the statistical significance among seroconversion rates across study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Qihan Li, Ph.D, Study Chair — Institude of Medical Biology, Chinese Academy of Medical Sciences; Jingsi Yang, Study Director — Institude of Medical Biology, Chinese Academy of Medical Sciences; Rongcheng Li, Principal Investigator — Guangxi Provincial Center for Disease Control and Prevention
Locations (1):
- Institute of Medical Biology -Chinese Academy of Medical Sciences Kunming, Yunnan, China 650118, Kunming, Yunnan, China